CLINICAL TRIAL: NCT01830738
Title: Laparoscopic Hysterectomy Via a Single Port, Peri-umbilical Technique Versus a Conventional Laparoscopic Technique : a Prospective, Randomized, Multicenter Study Evaluating the Length of Hospital Stay
Brief Title: Laparoscopic Hysterectomy Via a Single Port, Peri-umbilical Technique Versus a Conventional Laparoscopic Technique
Acronym: HOT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inclusion curve too poor.
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LOCAL/2012/VL-03; 2012-A01054-36 (Other: RCB number)
Record Dates: First submitted 2013-04-10; First posted 2013-04-12 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Hysterectomy
Keywords: laparoscopy; hysterectomy; single-port trocar; surgical technique; trocar

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peri-umbilical single-port (Experimental): Patients in this arm have a hysterectomy via a single-port peri-umbilical laparoscopic surgical technique.
  Intervention: Single-port, peri-umbilical hysterectomy
  Interventions: Procedure: Single-port, peri-umbilical hysterectomy
- Multi-port (Active Comparator): Patients in this arm have a hysterectomy via a conventional multi-port laparoscopic surgical technique.
  Intervention: Multi-port hysterectomy
  Interventions: Procedure: Multi-port hysterectomy

INTERVENTIONS:
Procedure: Single-port, peri-umbilical hysterectomy — Patients in this arm have a hysterectomy via a single-port peri-umbilical laparoscopic surgical technique.
  Arms: Peri-umbilical single-port
Procedure: Multi-port hysterectomy — Patients in this arm have a hysterectomy via a conventional multi-port laparoscopic surgical technique.
  Arms: Multi-port

SUMMARY:
The main objective of the study is the comparison of the effective duration of hospitalization following laparoscopic hysterectomy via a single-port peri-umbilical technique versus an conventional multi-port technique.

DETAILED DESCRIPTION:
The secondary objectives are to compare the following between the two arms of the study:

1. the difference between the real discharge date and the theoretical discharge date
2. measures related to intraoperative bleeding
3. operating time
4. postoperative pain
5. quality of life
6. abdominal wall complication rates
7. rates of further surgery and rehospitalization
8. use of material resources in the operating room
9. average costs of hospital stay
10. Costs of rehospitalization at 1 year
11. Indirect costs

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 12 months of follow-up
* The patient is declared fit by the anesthetist for an intervention by laparoscopy

Exclusion Criteria:

* The patient is not available for 12 months of follow-up
* The patient is participating in another study or is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient is not insured or beneficiary of a health insurance plan
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient cannot read French
* Patient with a history of pelvic radiotherapy
* Patient with a history of pelvic surgery or serious risk of major adhesions
* The patient is pregnant
* Contraindications for anesthesia for either surgical technique
* Promontofixation or lymphadenectomy
* No associated procedure other than morcellation or vaginal suture for extracting the hysterectomy specimen, unilateral or bilateral oophorectomy
* The patient has a known or suspected allergy to polyurethane
* Extended hysterectomy for neoplastic disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-02; Primary Completion 2014-08 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay in hours | Maximum 1 month (usually 3 to 5 days)

SECONDARY OUTCOMES:
Difference in hours between real discharge time and theoretical discharge time | 4 weeks
  Criteria for theoretical hospital discharge:
  * Visual analog scale for pain < 2 under stage 1 antalgics
  * No nausea, no vomiting
  * Resumption of transit, liquid and solid food
  * Capable of getting up, moving and going to the bathroom alone
  * Apyrexia
Bleeding/fluid loss: Difference between lavage fluids and aspiration fluids | Day 0 (during surgery)
Change in hemoglobin measure | Day 3 versus baseline
Change in hematocrit measure | Day 3 versus baseline
Surgical time, from first incision to closing | Day 0 (during surgery)
Visual analog scale for pain | 2 hours after end of surgery (Day 0)
Visual analog scale for pain | 3 times per day during hospitalisation (expected maximum of 3 to 5 days)
Questionnaire SF 36 | baseline
  Quality of Life
Questionnaire SF 36 | 4 weeks
  Quality of Life
Complication rate | Day 1
  Includes: hematomas around trocar sites; localized care for trocar infection or hematoma; surgery for trocar site herniation
Complication rate | 4 weeks
  Includes: hematomas around trocar sites; localized care for trocar infection or hematoma; surgery for trocar site herniation
Complication rate | 12 months
  Includes: hematomas around trocar sites; localized care for trocar infection or hematoma; surgery for trocar site herniation
Re-intervention/hospitalisation rate | 12 months
Surgical conversion rate | Day 0 (during surgery)
Trocar site infection rate | 4 weeks
Presence/absence of complications according to Clavien scale | Day 1
Presence/absence of complications according to Clavien scale | 12 months
Inventory of reusable material in the operating room and related costs. | Day 0 (after surgery)
Estimatin of indirect costs | 4 weeks
Estimation of direct costs | 12 months
Questionnaire SF 36 | 12 months
  Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Letouzey, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (3):
- France (3):
  - APHM - Hôpital de la Conception, Marseille
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - CHU de Saint Etienne - Hôpital Nord, Saint-Priest-en-Jarez